CLINICAL TRIAL: NCT03036501
Title: Open-label Study Investigating the Excretion Balance, Pharmacokinetics and Metabolism of a Single Oral Dose of [14C]-Labeled RO7034067 in Healthy Male Subjects
Brief Title: A Study Investigating the Excretion Balance, Pharmacokinetics and Metabolism of a Single Oral Dose of [14C]-Labeled Risdiplam (RO7034067) in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP39122; 2016-003461-26 (EudraCT Number)
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [^14C]-Risdiplam (Experimental): Participants will be administered with [^14C]-Risdiplam solution orally under fasted conditions on Day 1.
  Interventions: Drug: [^14C]-Risdiplam

INTERVENTIONS:
Drug: [^14C]-Risdiplam — [^14C]-Risdiplam 18 mg oral solution with approximately 0.75 megabecquerel MBq (20 microcuries [μCi]) of [14C]-labeled Risdiplam.

SUMMARY:
This is an open-label, non-randomized study investigating the excretion balance, PK and metabolism of a single oral dose of [14C]-labeled Risdiplam (RO7034067) in healthy male participants. This study will assess the characterize mass balance, routes and rates of elimination of [14C]-labeled Risdiplam (RO7034067), using conventional analytical methods and assess the pharmacokinetics of total drug related [14C]-radioactivity, Risdiplam (RO7034067) and its metabolite(s).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants, 35 to 65 years of age (inclusive)
* A body mass index between 18 to 30 kg/m^2 inclusive
* Agreement to use two methods of contraception, during the treatment period and for at least 4 months after the last dose of study drug. One of the contraceptive methods must be a condom. The second contraceptive method must include one of the following: diaphragm or cervical cap, intra-uterine device or system, or oral, injected or implanted hormonal method of contraception.
* No intention of donating sperm within 4 months of study drug administration
* Able to participate and willing to give written informed consent and to comply with the study requirements and restrictions
* Fluent in the language of the Investigator and study staff and able to communicate with the study staff

Exclusion Criteria:

* Any condition or disease detected during the medical interview/physical examination that would render the participant unsuitable for the study, place the participant at undue risk or interfere with the ability of the participant to complete the study in the opinion of the Investigator
* History of any clinically significant gastrointestinal, renal, hepatic, broncho- pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological or allergic disease, metabolic disorder, hypofertility, cancer or cirrhosis
* Participants with any clinically significant eye pathology affecting best-corrected visual acuity, or optic neuritis retinal abnormalities on spectral domain - optical coherence tomography and 7-field fundus color photography as assessed by an ophthalmologist
* History or evidence of (neuro) muscular disorders
* History or evidence of any medical condition potentially altering the absorption, metabolism or elimination of drugs. Surgical history of the gastrointestinal tract affecting gastric motility or altering the gastrointestinal tract
* History or evidence of skin disorders, as assessed by a thorough skin examination of the whole body
* History of malignancy in the past 5 years
* A history of clinically significant hypersensitivity (e.g., drugs, excipients) or allergic reactions
* Participants who, in the Investigator's judgment, pose a suicidal or homicidal risk, or any participant with a history of suicidal or homicidal attempts
* Any major illness within one month before the screening examination or any febrile illness within one week prior to screening and up to study drug administration
* History or presence of clinically significant ECG abnormalities before study drug administration or cardiovascular disease
* Clinically significant abnormalities in laboratory test results
* Positive results on tests for human immunodeficiency virus (HIV)-1 or HIV-2, hepatitis C virus or hepatitis B virus
* Any suspicion or history of alcohol abuse and/or suspicion of regular consumption of drugs of abuse
* Confirmed systolic blood pressure (SBP) greater than 150 or less than 90 mmHg, and diastolic blood pressure (DBP) greater than 95 or less than 50 mmHg
* Confirmed (based on the average of at least 3 consecutive measurements) resting pulse rate greater than 100 or less than 40 bpm
* Participation in an investigational drug or device study within 90 days prior to screening, as calculated from the day of follow-up from the previous study
* Smokers who regularly smoke more than 10 cigarettes daily or equivalent tobacco- containing products
* Dietary restrictions that would prohibit the consumption of standardized meals
* Use of any prohibited medications and food before study start and during the study
* Participants under judicial supervision, guardianship or curatorship
* Infrequent bowel movements (less than once per 24 hours on average)
* Regular work with ionizing radiation or radioactive material
* Participants who plan to attempt to father children within 4 months after study drug administration

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Dose Recovered as Total [14C]-radioactivity in Urine | Day 1 to Day 36
Cumulative Urinary Amount of Total [14C]-Radioactivity in Urine | Day 1 to Day 36
Percentage of Dose Recovered as Total [14C]-radioactivity in Feces | Day 1 to Day 36
Maximum Observed Plasma Concentration (Cmax) of Risdiplam | Day 1 to Day 36
Time to Maximum Observed Plasma Concentration of Risdiplam (Tmax) | Day 1 to Day 36
Area Under the Plasma Concentration-time Curve from Time 0 to Last Measurable Concentration Time Point (AUC0-last) | Day 1 to Day 36
Area Under Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) | Day 1 to Day 36
Apparent Terminal Elimination Half-Life (t1/2) | Day 1 to Day 36

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | Up to 10 weeks
Percentage of Participants with Laboratory, ECGs, Ophthalmological Assessments, And Vital Signs Abnormalities | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Pra International Group B.V, Groningen, Netherlands